CLINICAL TRIAL: NCT02947776
Title: Adjustment Post Stroke and Aphasia: Supporting Psychological Wellbeing Through Peer Befriending
Brief Title: Adjustment With Aphasia After Stroke: SUPERB
Acronym: SUPERB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Staff/16-17/06
Record Dates: First submitted 2016-10-13; First posted 2016-10-28 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-01

CONDITIONS: Stroke; Aphasia
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- USUAL (Active Comparator): Usual care
  Interventions: Behavioral: USUAL
- PEER (Experimental): Usual care + peer-befriending
  Interventions: Behavioral: PEER; Behavioral: USUAL

INTERVENTIONS:
Behavioral: PEER — The experimental group will receive usual care + peer befriending. Peer befriending aims to utilise the skills and 'lived experience' of people with longer-term aphasia to offer support to others with aphasia, starting at a time of transition (discharge from hospital and withdrawal of intensive therapeutic input) and increased need. It aims to help people develop their own strategies for adjusting to life post-stroke. Peer-befrienders will visit participants 6 times over a period of 3 months (+2 times within the next 6 months). The schedule, nature of visits, and goals (e.g. discuss concerns; pursue activities) will be agreed between the pair. Visits may include: conversation, problem solving, trips out, joint activities.
  Arms: PEER
Behavioral: USUAL — The control group will receive usual care, i.e. all health, social care and voluntary services available to them in their borough. It is not known what exactly usual care comprises for people with aphasia who are discharged in the community with low levels of psychological problems, and this project will help to document this.

SUMMARY:
Aims: This exploratory trial will:

1. Explore the feasibility of a definitive/phase III RCT on clinical and cost-effectiveness of peer-befriending for people with aphasia post-stroke.
2. Investigate psychological and social wellbeing outcomes of participants, significant others, and peer befrienders.
3. Explore the feasibility of a full economic evaluation of usual care + peer befriending versus usual care control.

Design: Single blind, mixed methods, parallel group phase II RCT comparing usual care + peer-befriending vs. usual care, starting at discharge from hospital. The study will deliver on four work packages: development phase; RCT; qualitative study; economic evaluation. Participants (n=60) will be assessed three times up to 10 months post-randomisation.

Outcome measures: Feasibility: feasibility of recruitment to definitive trial (proportion screened who meet criteria; proportion who consent; rate of consent); participant, significant other, peer befriender views on acceptability of procedures (qualitative study); number of missing/incomplete data on outcome measures; attrition rate at follow-up; potential value of conducting main trial using value of information analysis (economic evaluation); description of usual care; treatment fidelity of peer-befriending. Patient-reported outcomes will include mood, wellbeing, communication and social participation.

Benefits: Peer befriending may help avert some of the serious psychological consequences of stroke, and prevent the need for more complex and costly psychological therapies.

DETAILED DESCRIPTION:
Background: Stroke and aphasia can have a profound impact on people's lives. Depression is a common sequel of stroke, with rates remaining high even one year after stroke at 33%. It is associated with worse rehabilitation outcomes, increased carer strain, increased healthcare utilisation, and higher mortality. A recent audit of clinical psychology services for people with mood problems post-stroke across 10 UK stroke services found that the most common outcome of mood assessment was monitoring and advice, with less than half of patients with low mood receiving psychological intervention. There is a pressing need to evaluate systematically interventions that aim to improve psychosocial wellbeing for people with stroke and aphasia.

Aims: SUPERB trial aims to evaluate the feasibility of a phase III trial on the clinical and cost-effectiveness of a stepped care model level 1 intervention, peer befriending, for people with aphasia. Specifically it will:

1. Explore the feasibility of a definitive phase III randomised control trial (RCT) based on a) feasibility of recruitment and retention to the trial, b) acceptability of research procedures and outcome measures, c) acceptability of usual care + peer befriending vs. usual care control to participants, their significant others and peer support workers, d) documentation of usual care, e) treatment fidelity of peer befriending.
2. Explore psychological and social well-being outcomes as outcomes in a definitive trial for a) people with aphasia receiving usual care + peer befriending versus usual care control, b) their significant others, and c) peer befrienders.
3. Explore the feasibility of a full economic evaluation of usual care + peer befriending versus usual care control in a phase III RCT.

Intervention to be tested: The intervention group will receive peer befriending from stroke survivors with long-term aphasia who will be trained as peer befrienders. They will visit participants who have had a stroke more recently 6 times over a period of 3 months. An further 2 visits within the next 6 months will also be offered for a gradual transition to the end of the peer befriending. The schedule and nature of visits will be agreed between the pair at their first meeting. This meeting will also identify possible goals for the intervention e.g. to offer conversation, help with problem solving and social activities.

Methods: The overall study will last 3½ years and comprise a development phase (year 1) and a phase II RCT (years 2-3). The development phase will inform the intervention manual, the choice of outcome measures, fidelity practices and topic guides for participant interviews. This phase will be informed through a series of six workshops attended by six people with aphasia with experience of peer befriending. This will be followed by a pilot of the intervention, fidelity checking and all associated processes with 8 participants comparing usual care (n=4) with usual care + peer befriending (n=4).

The phase II RCT will be a single blind, mixed methods, parallel group design comparing usual care (n=30) with usual care + peer befriending (n=30) for people with aphasia post-stroke and low levels of psychological problems. Assessments and outcome measures for participants and significant others will be administered before randomisation with outcome measures re-administered at 4 and 10 months post-randomisation. Peer befrienders will complete outcome measures before training and after they have completed the visits for two participants. In addition, this RCT will include a qualitative study and a feasibility economic evaluation. The qualitative study will use semi-structured interviews of purposively sampled participants (n=20) and significant others (n=10) from both arms of the trial, and peer befrienders. The feasibility economic evaluation will utilise the EQ-5D and a stroke-adapted version of the CSRI.

Outcomes: RCT: feasibility of recruitment of participants to definitive trial (including proportion screened who meet criteria; proportion who consent; rate of consent); number of missing/incomplete data on outcome measures; attrition rate at follow-up; potential value of conducting main trial using value of information analysis (economic evaluation); description of usual care; treatment fidelity of peer befriending. Patient-reported outcomes will include mood, wellbeing, communication and social participation. Qualitative study: participant, significant other, peer befriender views on acceptability of procedures and experiences of care received. Economic evaluation: cost outcomes, average costs, costs per participant and mean difference between trial arms, description of resources used and overall cost effectiveness.

Benefits: This study will inform on whether peer befriending is a suitable intervention to explore further, in terms of averting some of the serious psychological consequences of stroke, and preventing the need for more complex and costly psychological therapies.

ELIGIBILITY:
Inclusion Criteria:

Participants with aphasia:

* Over 18;
* Fluent premorbid users of English (confirmed by relative or self report);
* Presence of aphasia due to stroke; and
* Low levels of emotional distress (score of ≤2 on Depression Intensity Scale Circles). The latter will ensure that they do not require immediate level 2 or 3 psychological input. People who score 2 (which is also the median on DISCS) and who the MDT deems do not need stepping up or stepping up is not available, will still be eligible to take part.

Significant Others: each participant with aphasia will nominate one significant other, who is their closest confidant and who is over 18 years of age. If participants live alone their significant other should be someone that they see at least once a week.

Peer befrienders: will be people with mild-moderate aphasia (score score a minimum 5/10 for auditory comprehension and 5/10 for verbal expression in the Frenchay Aphasia Screening Test) who are over 18 years of age, are at least one year post-stroke

Exclusion Criteria:

Participants will be excluded if they have:

* Other diagnoses affecting cognition or mental health (based on medical records for participants with aphasia and self-report for significant others and peer befrienders, as well as the GHQ-12 as a depression screen for peer befrienders: will be excluded if they score 3 or more);
* Severe uncorrected visual or hearing problems (based on medical records for participants with aphasia and self-report for significant others and peer befrienders);
* Severe or potentially terminal co-morbidities, on grounds of frailty (based on medical records for participants with aphasia and self-report for significant others and peer befrienders).

Participants with aphasia will also be excluded if they are:

• Discharged to a geographical location outside the borough of the recruiting hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
General Health Questionnaire-12 (GHQ-12) continuous total score | 4 months post randomisation
  For participants with aphasia.
Depression Intensity Scale Circles (DISCS) continuous total score | 4 months post randomisation
  The DISCS will be treated as the primary outcome measure only if there is ≥10% missing data in the GHQ-12 due to severity of aphasia, otherwise it will be a secondary outcome measure.
General Health Questionnaire-12 (GHQ-12) continuous total score | 10 months post randomisation
  For participants with aphasia.
Depression Intensity Scale Circles (DISCS) continuous total score | 10 months post randomisation
  The DISCS will be treated as the primary outcome measure only if there is ≥10% missing data in the GHQ-12 due to severity of aphasia, otherwise it will be a secondary outcome measure.

SECONDARY OUTCOMES:
Short Warwick Edinburgh Mental Well-being Scale (SWEMWBS) continuous total score. | 4 months post randomisation
  For participants with aphasia.
Short Warwick Edinburgh Mental Well-being Scale (SWEMWBS) continuous total score. | 10 months post randomisation
  For participants with aphasia.
Communicative Participation Item Bank (CPIB) continuous total score | 4 months post randomisation
  For participants with aphasia.
Communicative Participation Item Bank (CPIB) continuous total score | 10 months post randomisation
  For participants with aphasia.
Community Integration Questionnaire (CIQ) continuous total score | 4 months post randomisation
  For participants with aphasia.
Community Integration Questionnaire (CIQ) continuous total score | 10 months post randomisation
  For participants with aphasia.
Proportion with high emotional distress vs low emotional distress as measured using the GHQ-12 (high distress = score of 3 or more, low distress = score of 0-2) | 4 months post randomisation
  For participants with aphasia.
Proportion with high emotional distress vs low emotional distress as measured using the GHQ-12 (high distress = score of 3 or more, low distress = score of 0-2) | 10 months post randomisation
  For participants with aphasia.
Warwick Edinburgh Mental Well-being Scale (WEMWBS) continuous total score | 4 months post randomisation
  For significant others.
Warwick Edinburgh Mental Well-being Scale (WEMWBS) continuous total score | 10 months post randomisation
  For significant others.
General Health Questionnaire-28 (GHQ-28) continuous total score. The GHQ-28 also provides four subscale scores (somatic symptoms, anxiety/insomnia, severe depression, and social dysfunction), which will be looked at descriptively. | 4 months post randomisation
  For significant others.
General Health Questionnaire-28 (GHQ-28) continuous total score. The GHQ-28 also provides four subscale scores (somatic symptoms, anxiety/insomnia, severe depression, and social dysfunction), which will be looked at descriptively. | 10 months post randomisation
  For significant others.
Bakas Caregiving Outcome Scale (BCOS) continuous total score | 4 months post randomisation
  For significant others.
Bakas Caregiving Outcome Scale (BCOS) continuous total score | 10 months post randomisation
  For significant others.
Warwick Edinburgh Mental Well-being Scale (WEMWBS) continuous total score | ~ 6 months
  For peer befrienders. Outcomes will be assessed on completion of 2 befriending cycles
Community Integration Questionnaire (CIQ) continuous total score | ~ 6 months
  For peer befrienders. Outcomes will be assessed on completion of 2 befriending cycles

OTHER OUTCOMES:
Communication Confidence Rating Scale for people with aphasia (CCRSA) | 4 months post randomisation
  Exploratory measure for participants with aphasia.
Communication Confidence Rating Scale for people with aphasia (CCRSA) | 10 months post randomisation
  Exploratory measure for participants with aphasia.
Friendship Scale (FS) | 4 months post randomisation
  Exploratory measure for participants with aphasia.
Friendship Scale (FS) | 10 months post randomisation
  Exploratory measure for participants with aphasia.
EQ-5D-5L | 4 months post randomisation
  Economic evaluation outcome.
EQ-5D-5L | 10 months post randomisation
  Economic evaluation outcome.
Stroke adapted Client Service Receipt Inventory (CSRI) | 4 months post randomisation
  Economic evaluation outcome.
Stroke adapted Client Service Receipt Inventory (CSRI) | 10 months post randomisation
  Economic evaluation outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Hilari, Principal Investigator — City, University of London
Locations (5):
- United Kingdom (5):
  - The Royal London Hospital, London
  - Homerton University Hospital, London
  - University College London Hospital, London
  - The Royal Free Hospital, London
  - The National Hospital for Neurology and Neurosurgery, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data may be shared e.g. for meta-analyses

REFERENCES:
- [Background] Hilari K, Behn N, Marshall J, Simpson A, Thomas S, Northcott S, Flood C, McVicker S, Jofre-Bonet M, Moss B, James K, Goldsmith K. Adjustment with aphasia after stroke: study protocol for a pilot feasibility randomised controlled trial for SUpporting wellbeing through PEeR Befriending (SUPERB). Pilot Feasibility Stud. 2019 Jan 22;5:14. doi: 10.1186/s40814-019-0397-6. eCollection 2019. PMID 30693094
- [Derived] Behn N, Moss B, McVicker S, Roper A, Northcott S, Marshall J, Thomas S, Simpson A, Flood C, James K, Goldsmith K, Hilari K. SUpporting wellbeing through PEeR-Befriending (SUPERB) feasibility trial: fidelity of peer-befriending for people with aphasia. BMJ Open. 2021 Aug 2;11(8):e047994. doi: 10.1136/bmjopen-2020-047994. PMID 34341046
- [Derived] Moss B, Behn N, Northcott S, Monnelly K, Marshall J, Simpson A, Thomas S, McVicker S, Goldsmith K, Flood C, Hilari K. "Loneliness can also kill:" a qualitative exploration of outcomes and experiences of the SUPERB peer-befriending scheme for people with aphasia and their significant others. Disabil Rehabil. 2022 Sep;44(18):5015-5024. doi: 10.1080/09638288.2021.1922519. Epub 2021 Jun 4. PMID 34086521
- [Derived] Northcott S, Behn N, Monnelly K, Moss B, Marshall J, Thomas S, Simpson A, McVicker S, Flood C, Goldsmith K, Hilari K. "For them and for me": a qualitative exploration of peer befrienders' experiences supporting people with aphasia in the SUPERB feasibility trial. Disabil Rehabil. 2022 Sep;44(18):5025-5037. doi: 10.1080/09638288.2021.1922520. Epub 2021 May 23. PMID 34027757
- [Derived] Hilari K, Behn N, James K, Northcott S, Marshall J, Thomas S, Simpson A, Moss B, Flood C, McVicker S, Goldsmith K. Supporting wellbeing through peer-befriending (SUPERB) for people with aphasia: A feasibility randomised controlled trial. Clin Rehabil. 2021 Aug;35(8):1151-1163. doi: 10.1177/0269215521995671. Epub 2021 Feb 24. PMID 33624514
- See also: Full text of SUPERB protocol paper available on link above — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-019-0397-6